CLINICAL TRIAL: NCT02476552
Title: Absorption, Metabolism, Excretion, and the Determination of Absolute Bioavailability of Niraparib in Subjects With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-30-5015-C
Record Dates: First submitted 2015-05-29; First posted 2015-06-19 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — niraparib; Product Labeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Niraparib Oral and IV (Experimental): Single Oral dose of Niraparib capsules (unlabeled active pharmaceutical ingredient) orally and a 15-minute IV infusion of Niraparib (labeled active pharmaceutical ingredient)
  Interventions: Drug: Niraparib IV (Labeled); Drug: Niraparib Oral Capsules (Unlabeled)
- Niraparib Oral (Experimental): Single Oral dose of Niraparib capsules (labeled active pharmaceutical ingredient)
  Interventions: Drug: Niraparib Oral Capsules (Labeled)

INTERVENTIONS:
Drug: Niraparib Oral Capsules (Labeled) — Single 300 mg dose of niraparib
  Arms: Niraparib Oral
Drug: Niraparib IV (Labeled) — Intravenous (IV) infusion of 100 μg niraparib (containing approximately 1 μCi of [14C]-niraparib)
  Arms: Niraparib Oral and IV
Drug: Niraparib Oral Capsules (Unlabeled) — Single 300 mg dose of niraparib (unlabeled active pharmaceutical ingredient)
  Arms: Niraparib Oral and IV

SUMMARY:
This is an open-label study with 2 parts, plus an extension study following completion of Parts 1 or 2, that is being conducted in approximately 12 subjects (6 subjects in Part 1; 6 subjects in Part 2) with cancer to examine the absorption, metabolism, excretion, and absolute bioavailability of niraparib.

DETAILED DESCRIPTION:
Part 1: After an overnight fast of at least 10 hours, subjects will receive a single, oral dose of niraparib (unlabeled active pharmaceutical ingredient) on Day 1. Two hours after the oral dose, subjects will receive a 15-minute IV infusion of niraparib (labeled pharmaceutical ingredient).

Part 2: After an overnight fast of at least 10 hours, subjects will receive a single, oral dose of niraparib, labeled active pharmaceutical ingredient.

ELIGIBILITY:
Inclusion Criteria:

* Subject, male or female, is at least 18 years of age.
* Subject has histologically or cytologically confirmed diagnosis of metastatic or locally advanced solid tumors that have failed to respond to standard therapy, have progressed despite standard therapy, refuse standard therapy, or for which no standard therapy exists, and that may benefit from treatment with a poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) inhibitor. The diagnosis must be confirmed with a previous computed tomography (CT) scan.
* The subject has adequate organ function:
* Subject must have an ECOG performance status of 0 to 2.
* Female subjects of childbearing potential must have a negative serum pregnancy test (beta human chorionic gonadotropin [hCG]) within 72 hours prior to receiving the first dose of study drug.

Exclusion Criteria:

* Subject has undergone palliative radiotherapy within 1 week of study drug administration, encompassing >20% of the bone marrow.
* Subject has persistent >Grade 2 toxicity from prior cancer therapy.
* Subject has known hypersensitivity to the components of niraparib.
* Subject has had major surgery within 3 weeks of study drug administration or has not recovered from all effects of any major surgery.
* Subject is considered a medical risk due to a serious, uncontrolled medical disorder; nonmalignant systemic disease; or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days of the Screening Visit) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent.
* Subject has participated in a radioactive clinical study and has received an investigational radiolabeled drug within 6 months prior to study drug administration (for subjects participating in Part 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Oral bioavailability (F) will be derived using F=AUCoral / AUCiv as a % | 0 - 22 days
  Absolute bioavailability of niraparib will be calculated as the ratio of dose normalized oral to IV niraparib exposure

SECONDARY OUTCOMES:
AUC0-last | 0 - 22 days
  AUC (Area Under the Curve) from time 0 to the last quantifiable concentration
Cmax | 0 - 22 days
  Observed Maximum plasma Concentration

CONTACTS AND LOCATIONS:
Overall Officials: Shefali Agarwal, MD, Study Director — Tesaro, Inc.
Locations (1):
- The Netherlands Cancer Institute, Amsterdam, Netherlands